CLINICAL TRIAL: NCT01967134
Title: Phase I Open Label Dose-Escalation Study to Evaluate the Safety and Immunogenicity of H56:IC31 (AERAS-456) in HIV-negative Adults With and Without Latent Tuberculosis Infection
Brief Title: Safety and Immunogenicity Study of AERAS-456 Vaccine for Tuberculosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeras (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: C-032-456
Record Dates: First submitted 2013-10-18; First posted 2013-10-22 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-06

CONDITIONS: Latent Tuberculosis; Latent Tuberculosis Bacteriology and Histology Unknown
Keywords: HIV Negative
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- H56:IC31 (50 ug H56) LTBI Neg (Experimental): LTBI Negative 3 Doses
  Interventions: Biological: H56:IC31
- H56:IC31 (15 ug H56) LTBI Pos (Experimental): LTBI Positive 3 Doses
  Interventions: Biological: H56:IC31
- H56:IC31 (50 ug H56) LTBI Pos (Experimental): LTBI Positive 3 Doses
  Interventions: Biological: H56:IC31

INTERVENTIONS:
Biological: H56:IC31 — H56:IC31 contains a fusion protein (referred to as H56 antigen, or H56) of 3 mycobacterial antigens (the early secreted antigens Ag85B and ESAT-6, and the latency antigen Rv2660c) formulated in the Th1-stimulating IC31 adjuvant.
  Other Names: AERAS 456

SUMMARY:
This is a Phase I, open-label, dose-escalation study with three study groups. This study will be conducted in 25 HIV negative subjects, 17 of whom will have Latent Tuberculosis Infection (LTBI) and 8 of whom will not have LTBI at study enrollment. The investigational product is AERAS-456 at a dose of 15 ug of H56 antigen with IC31 500 nmol KLK (15/500), and a dose of 50 ug of H56 antigen with IC31 500 nmol KLK (50/500). The vaccine is administered by intramuscular injection.

DETAILED DESCRIPTION:
This is a Phase I, open-label, dose-escalation study with three study groups. This study will be conducted in 25 HIV negative subjects, 17 of whom will have Latent Tuberculosis Infection (LTBI) and 8 of whom will not have LTBI at study enrollment. The investigational product is H56:IC31 (AERAS-456) at a dose of 15 ug of H56 antigen with IC31 500 nmol KLK (15/500), and a dose of 50 ug of H56 antigen with IC31 500 nmol KLK (50/500). The vaccine is administered by intramuscular (IM) injection.

Subjects will be assigned to a study group based on LTBI status at enrollment and time of completion of screening. Subjects without LTBI will be assigned to Group 1. Subjects with LTBI will be sequentially assigned to Groups 2 and 3 based on the order in which they complete screening. All subjects will receive a first dose of study vaccine on Study Day 0, a second dose of study vaccine on Study Day 56, and a third dose of study vaccine on Study Day 112. Enrollment of subjects into Group 2 will begin only after a review of safety data from the 14-day period after initial vaccination of all subjects in Group 1. Likewise, enrollment of subjects into Group 3 will begin only after the corresponding review of safety data from Group 2.

The total duration of study follow-up for all subjects is 210 days. Study groups 1-2 will enroll 8 subjects each and study group 3 will enroll 9 subjects. This study is planned at a single clinical site in South Africa. The sizes specified for each study group were selected because they are judged to be adequate for preliminary safety and immunogenicity evaluations for a Phase I study rather than for statistical reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Has completed the written informed consent process
2. Is male or female
3. Is aged 18 through 50 years on Study Day 0
4. Females: Ability to avoid pregnancy during the trial: Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must avoid pregnancy with an acceptable method of avoiding pregnancy from 28 days prior to administration of the study vaccine through the end of the study.
5. Has general good health, confirmed by medical history and physical examination
6. Is able and willing to complete the full follow-up period of 210 days as required by the protocol
7. Is able and willing to commit to avoiding elective surgery for the duration of the study
8. Is able and willing to stay in contact with the study site for the duration of the study
9. [Groups 2 & 3] Has latent tuberculosis infection (LTBI), diagnosed by a positive Quantiferon (QFT)
10. Has completed simultaneous enrollment in the Registry Protocol

Exclusion Criteria:

1. Axillary temperature 37.5 C
2. Abnormal laboratory values from blood collected within 7 days prior to Study Day 0 vaccination as follows:

   * hemoglobin, hematocrit, platelet count, absolute neutrophil count, or absolute lymphocyte count below lower limit of normal (LLN).
   * white blood cell count above upper limit of normal (ULN) or below LLN
   * alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, alkaline phosphatase (ALP), or creatinine above ULN.
3. Abnormal urinalysis that, in the opinion of the investigator, indicates systemic or local disease.
4. History or evidence of tuberculosis disease, including but not limited to pulmonary tuberculosis, pleural tuberculosis, lymph node tuberculosis or tuberculosis meningitis.
5. [Group 1] Evidence of latent tuberculosis infection (LTBI), defined as a positive screening QFT or a history of a positive TST or QFT.
6. Received a tuberculin skin test (TST) or bacillus Calmette-Guerin (BCG) within 45 days prior to Study Day 0.
7. Received investigational Mtb vaccine at any time prior to Study Day 0.
8. History or evidence of autoimmune disease.
9. History or laboratory evidence of HIV infection.
10. History or laboratory evidence of Hepatitis B or C.
11. Used immunosuppressive medication (other than inhaled or topical immunosuppressants) within 45 days prior to Study Day 0.
12. Received immunoglobulin or blood products within 45 days prior to Study Day 0
13. Received any investigational product within 45 days prior to Study Day 0, or plans to participate in any other study involving administration of investigational product during the study period.
14. Inability to discontinue daily medications, except contraceptives, inhaled or topical immunosuppressants, or nutritional supplements, during the study period.
15. Documented history of allergic reaction or hypersensitivity to any component of the study vaccine.
16. Female subjects: currently pregnant or lactating/nursing; or positive serum pregnancy test during screening; or positive urine pregnancy test on the day of Study Day 0, Study Day 56, or Study Day 112 vaccination.
17. History or evidence of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may compromise the safety of the subject in the study or interfere with the evaluation of the safety or immunogenicity of the vaccine.
18. History of dermatologic disease or skin features that, in the opinion of the investigator, may interfere with the assessment of injection site reactions.
19. History or evidence of any medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the subject will comply with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angelique Luabeya, MD, Principal Investigator — University of Cape Town South African Tuberculosis Vaccine Initiative
Locations (1):
- SATVI Project Office, Brewelskloof Hospital, Worcester, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luabeya AK, Kagina BM, Tameris MD, Geldenhuys H, Hoff ST, Shi Z, Kromann I, Hatherill M, Mahomed H, Hanekom WA, Andersen P, Scriba TJ; H56-032 Trial Study Group; Schoeman E, Krohn C, Day CL, Africa H, Makhethe L, Smit E, Brown Y, Suliman S, Hughes EJ, Bang P, Snowden MA, McClain B, Hussey GD. First-in-human trial of the post-exposure tuberculosis vaccine H56:IC31 in Mycobacterium tuberculosis infected and non-infected healthy adults. Vaccine. 2015 Aug 7;33(33):4130-40. doi: 10.1016/j.vaccine.2015.06.051. Epub 2015 Jun 19. PMID 26095509

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | H56:IC31 (50 ug H56) LTBI Neg | H56:IC31 (15 ug H56) LTBI Pos | H56:IC31 (50 ug H56) LTBI Pos
Started | 8 | 8 | 9
Completed | 8 | 7 | 9
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H56:IC31 (50 ug H56) LTBI Neg | H56:IC31 (15 ug H56) LTBI Pos | H56:IC31 (50 ug H56) LTBI Pos | Total
Number analyzed (Participants) | 8 | 8 | 9 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 9 | 25
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 5 | 15
  Male | 4 | 2 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 9 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 5
  White | 0 | 0 | 0 | 0
  More than one race | 5 | 7 | 8 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 8 | 8 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Adverse Event (AE) Through Day 210
Description: Solicited AEs: through 14 days after each vaccination Unsolicited AEs: post-vaccination on Study Days 0, 56, and 112 through 28 days after vaccination Injection site reactions and axillary lymphadenopathy: post-injection on the day of each vaccination, and Study Days 2 , 7, 14, and 28 days after each vaccination Serious adverse events (SAE): through Study Day 210
Time Frame: Through Study Day 210
Population: Safety population
Measure: Number; unit: Participants
Arm/Group | H56:IC31 (50 ug H56) LTBI Neg | H56:IC31 (15 ug H56) LTBI Pos | H56:IC31 (50 ug H56) LTBI Pos
Number analyzed (Participants) | 8 | 8 | 9
Participants
  Participants with at least one AE after any dose | 8 | 8 | 9
  Participants with at least one AE after 3rd dose | 6 | 7 | 4

2. Secondary Outcome: Median % Change in Response to Peptides From Vaccine Antigen Ag85B From Pre-vaccination to Day 70 in Participants Who Received Two Vaccinations
Description: Whole blood ICS Percent Antigen-Specific T Cell UNS-subtracted Cytokine Response Antigen: Ag85B Cytokine(s): G+2+17+T+
  %CD4+ T Cell Response
Time Frame: Study Day 70
Population: All vaccinated subjects
Measure: Median (95% Confidence Interval); unit: % change from pre-vacc to day 70
Arm/Group | H56:IC31 (50 ug H56) LTBI Neg | H56:IC31 (15 ug H56) LTBI Pos | H56:IC31 (50 ug H56) LTBI Pos
Number analyzed (Participants) | 8 | 8 | 9
% change from pre-vacc to day 70 | 0.0008 [-0.0002 to 0.0026] | 0.0050 [0.0016 to 0.0075] | 0.0019 [0.0011 to 0.0044]

3. Secondary Outcome: Median % Change in Response to Peptides From Vaccine Antigen ESAT-6 From Pre-vaccination to Day 70 in Participants Who Received Two Vaccinations
Description: Percent Antigen-Specific T Cell UNS-subtracted Cytokine Response 12-Hour Whole Blood Intracellular Cytokine Staining (ICS) Assay Antigen: ESAT6 Cytokine(s): G+2+17+T+
  %CD4+ T Cell Response
Time Frame: Study Day 70
Population: All vaccinated subjects
Measure: Median (95% Confidence Interval); unit: % change from pre-vacc to day 70
Arm/Group | H56:IC31 (50 ug H56) LTBI Neg | H56:IC31 (15 ug H56) LTBI Pos | H56:IC31 (50 ug H56) LTBI Pos
Number analyzed (Participants) | 8 | 8 | 9
% change from pre-vacc to day 70 | 0.0000 [0.0000 to -0.0003] | 0.0005 [0.0001 to 0.0009] | 0.0005 [0.0000 to 0.0012]

4. Secondary Outcome: Number of Participants Who Received at Least Two Vaccinations and Tested Positive for Mtb Infection on Day 210
Description: Measure of Mtb positivity by QuantiFERON-TB Gold In-Tube Number of Positive Responses and Shift from Screening to Study Day 210 Post-Vaccination Responses
Time Frame: Study Day 210
Population: All vaccinated subjects
Measure: Count of Participants; unit: Participants
Arm/Group | H56:IC31 (50 ug H56) LTBI Neg | H56:IC31 (15 ug H56) LTBI Pos | H56:IC31 (50 ug H56) LTBI Pos
Number analyzed (Participants) | 8 | 8 | 9
Participants | 2 | 6 | 9

5. Secondary Outcome: Median % Change in Response to Peptides From Vaccine Antigen Ag85AB From Pre-vacc to Day 210
Description: Responses to vaccine antigen Ag85B measure by Interferon gamma (IFN-γ) ELISpot assay Unstimulated-subtracted IFN-γ ELISpot Response (Spot forming units/10^6 PBMC) Antigen: Ag85B
Time Frame: Study Day 210
Population: Subjects in all vaccinated population with available data
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | H56:IC31 (50 ug H56) LTBI Neg | H56:IC31 (15 ug H56) LTBI Pos | H56:IC31 (50 ug H56) LTBI Pos
Number analyzed (Participants) | 7 | 1 | 7
percent change | 36.6667 [-4.9916 to 83.0868] | -8.3333 [NA to NA] — n=1 | 80.0000 [11.6905 to 164.9762]

ADVERSE EVENTS:
Time Frame: Solicited AEs: Thru 14 days after each vaccination Unsolicited AEs: 28 days after each vaccination SAEs: Days 0-210
Groups:
- Aeras-456 (50 ug H56/500 Nmol IC31) LTBI Negative: LTBI Negative 3 Doses
  Aeras-456: H56:IC31 (designated as AERAS-456 for Aeras-sponsored clinical development) contains a fusion protein (referred to as H56 antigen, or H56) of 3 mycobacterial antigens (the early secreted antigens Ag85B and ESAT-6, and the latency antigen Rv2660c) formulated in the Th1-stimulating IC31 adjuvant.
- Aeras-456 (15 ug H56/500 Nmol IC31) LTBI Positive; Aeras-456 (50 ug H56 / 500 Nmol IC31) LTBI Positive: LTBI Positive 3 Doses
  Aeras-456: H56:IC31 (designated as AERAS-456 for Aeras-sponsored clinical development) contains a fusion protein (referred to as H56 antigen, or H56) of 3 mycobacterial antigens (the early secreted antigens Ag85B and ESAT-6, and the latency antigen Rv2660c) formulated in the Th1-stimulating IC31 adjuvant.
Arm/Group | Aeras-456 (50 ug H56/500 Nmol IC31) LTBI Negative | Aeras-456 (15 ug H56/500 Nmol IC31) LTBI Positive | Aeras-456 (50 ug H56 / 500 Nmol IC31) LTBI Positive
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aeras-456 (50 ug H56/500 Nmol IC31) LTBI Negative (N=8) | Aeras-456 (15 ug H56/500 Nmol IC31) LTBI Positive (N=8) | Aeras-456 (50 ug H56 / 500 Nmol IC31) LTBI Positive (N=9)
Bradycardia (Cardiac disorders) | 4 (5) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (7) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (9) | 4 (8) | 2 (3)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 5 (12) | 7 (18) | 6 (11)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 2 (2) | 4 (5)
Injection site warmth (General disorders) | 5 (9) | 6 (10) | 6 (10)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 2 (3) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (5) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (2) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Protein urine (Investigations) | 5 (6) | 0 (0) | 0 (0)
Red blood cells urine (Investigations) | 2 (2) | 2 (2) | 2 (2)
White blood cell count increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (7) | 1 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (10) | 2 (5) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (4) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No